CLINICAL TRIAL: NCT03985423
Title: A Phase 2/3, Open-label, Single Arm, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Emapalumab in Adult Patients With Hemophagocytic Lymphohistiocytosis
Brief Title: A Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Emapalumab in Adult Patients With HLH
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Light Chain Bioscience - Novimmune SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NI-0501-10
Record Dates: First submitted 2019-05-23; First posted 2019-06-13 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Hemophagocytic Lymphohistiocytoses
Keywords: interferon gamma; emapalumab; adult HLH; malignancy-associated HLH; CXCL9
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Emapalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Emapalumab (Experimental): Patients were administered Emapalumab-Lzsg by intravenous (i.v.) infusion over a period of 1 to 2 hours, at an initial dose of 6 mg/kg and continued at 3 mg/kg, every 3 days for the first 2 weeks (Study Day [SD] 15), and then twice-a-week. If the treating physician deemed appropriate, the dose of emapalumab could be increased (up to 10 mg/kg), guided by clinical and laboratory response.
  Interventions: Drug: Emapalumab-Lzsg

INTERVENTIONS:
Drug: Emapalumab-Lzsg — Patients were administered Emapalumab-Lzsg by intravenous (i.v.) infusion over a period of 1 to 2 hours, at an initial dose of 6 mg/kg and continued at 3 mg/kg, every 3 days for the first 2 weeks (Study Day [SD] 15), and then twice-a-week. If the treating physician deemed appropriate, the dose of emapalumab could be increased (up to 10 mg/kg), guided by clinical and laboratory response.
  Other Names: NI-0501

SUMMARY:
Hemophagocytic lymphohistiocytosis (HLH) is a rare, life-threatening condition characterized by uncontrolled hyperinflammation which may develop on the background of several clinical conditions (e.g. autoimmune disease, infection, malignancy). Emapalumab (previously referred to as NI-0501) is a monoclonal antibody neutralizing interferon-gamma (IFN-gamma), a key cytokine driving the inflammation and tissue damage seen in HLH. The purpose of this study is to assess the efficacy, safety and pharmacokinetics of emapalumab in adult patients with secondary HLH.

DETAILED DESCRIPTION:
Study NI-0501-10 is an open-label, single arm, multicenter, Phase 2/3 interventional study.

The study enrolls adult patients with hemophagocytic lymphohistiocytosis (HLH), specifically newly diagnosed patients with malignancy-associated HLH (M-HLH), and newly diagnosed or previously treated patients with non-malignancy-associated HLH.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of age 18 and older at the time of HLH diagnosis
* Fulfilment of 5 of the 8 HLH-2004 clinical criteria
* Patients diagnosed with malignancy-associated HLH must be treatment naïve; patients diagnosed with HLH driven by any other etiology or idiopathic can be either treatment naïve or treatment experienced
* Patients with non-malignancy-associated or idiopathic HLH who have already received conventional therapy for HLH must have failed prior treatment as per the treating physician's judgement
* Informed consent signed by the patient or by the patient's legally authorized representative(s) (as required by local law)
* Willing to use highly effective methods of contraception from study drug initiation to 6 months after the last dose of study drug, if female and of childbearing potential.

Exclusion Criteria:

* Primary HLH
* Current or scheduled administration of therapies known to trigger the cytokine release syndrome (e.g. chimeric antigen receptor (CAR)-modified T cells, bispecific T cell-engaging antibodies)
* Current or scheduled administration of PD-1/PD-L1/CTLA-4 inhibitors
* Life-expectancy associated with the underlying disease (triggering HLH) < 3 months
* Ongoing participation in an investigational trial, or administration of any investigational treatment within 30 days
* History of hypersensitivity or allergy to any components of emapalumab
* Active mycobacteria, Histoplasma capsulatum, or Leishmania infections
* Evidence of latent tuberculosis
* Receipt of a bacille Calmette-Guerin (BCG) vaccine within 12 weeks prior to Screening
* Receipt of a live or attenuated live (other than BCG) vaccine within 6 weeks prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Radmila Kanceva, Study Director — Swedish Orphan Biovitrum
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2/3, open-label, single arm study was conducted in adult patients with hemophagocytic lymphohistiocytosis (HLH) at a single center in the United States of America.
Pre-assignment Details: The study consisted of a screening (up to 2 weeks), treatment period (until clinically satisfactory response was achieved), and follow-up period (1 year). A total of 7 patients were enrolled in the study and treated.
Groups:
- Emapalumab: Patients were administered emapalumab 6 milligram per kilogram (mg/kg) intravenous (IV) infusion for 1 to 2 hours, and continued at 3 mg/kg every 3 days for the first 2 weeks, and then twice-a-week until clinically satisfactory response was achieved.
  If the treating physician deemed appropriate, the dose of emapalumab could be increased (up to 10 mg/kg), guided by clinical and laboratory response.
Period: Overall Study
Arm/Group | Emapalumab
Started | 7
Completed | 0
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Death | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lack of insurance and citizenship | 1

BASELINE CHARACTERISTICS:
Population: The All Treated analysis set included all patients who received at least 1 dose or 1 incomplete dose of emapalumab.
Groups:
- Emapalumab: Patients were administered emapalumab 6 mg/kg IV infusion for 1 to 2 hours, and continued at 3 mg/kg every 3 days for the first 2 weeks, and then twice-a-week until clinically satisfactory response was achieved.
  If the treating physician deemed appropriate, the dose of emapalumab could be increased (up to 10 mg/kg), guided by clinical and laboratory response.
Arm/Group | Emapalumab
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (17.64)
Age, Continuous [Median (Full Range); unit: years] | 50 [25 to 73]
Age, Customized [Count of Participants; unit: Participants]
  >= 18 and 64 years | 6
  >= 65 and 84 years | 1
  >= 85 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 4
  Race: Other | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
Weight [Mean (Standard Deviation); unit: kg] | 80.84 (11.855)
Height [Mean (Standard Deviation); unit: centimeter] | 168.59 (12.234)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Achievement of either a Complete or Partial Response
  Complete Response is adjudicated if the following are observed:
  * No fever = body temperature <37.5°C
  * Normal spleen size
  * No cytopenia = Absolute Neutrophil Counts >=1.0x10^9/L and platelet count >=100x10^9/L [absence of G-CSF and transfusion support must be documented for at least 4 days to report no cytopenia]
  * No hyperferritinemia = serum level is <2000 µg/L
  * No evidence of coagulopathy, i.e., normal D-Dimer and/or normal (>150 mg/dL) fibrinogen levels
  * No neurological and CSF abnormalities attributed to HLH
  * No sustained worsening of sCD25 (as indicated by at least two consecutive measurements that are >2-fold higher than baseline)
  Partial Response is adjudicated if there is an improvement (>50% change from baseline or normalization) of at least 3 HLH clinical and laboratory criteria (including Central Nervous System abnormalities).
Time Frame: Week 4
Population: Since the study was prematurely terminated, no data was collected for the primary efficacy endpoint.
Arm/Group | Emapalumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Best Response on Treatment
Description: As no data are reported for this outcome measure, additional method is not applicable in the outcome measure description.
Time Frame: Week 4; End of Treatment Visit (on average of 12 weeks)
Population: Since the study was prematurely terminated, no data was collected for the secondary efficacy endpoints.
Arm/Group | Emapalumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Response
Description: as for outcome 2
Time Frame: End of Treatment Visit (on average of 12 weeks)
Population: Since the study was prematurely terminated, no data was collected for the secondary efficacy endpoints.
Arm/Group | Emapalumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: as for outcome 2
Time Frame: End of Treatment Visit (on average of 12 weeks)
Population: Since the study was prematurely terminated, no data was collected for the secondary efficacy endpoints.
Arm/Group | Emapalumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Complete Response or Partial Response
Description: as for outcome 2
Time Frame: Week 4; End of Treatment visit (on average of 12 weeks)
Population: Since the study was prematurely terminated, no data was collected for the secondary efficacy endpoints.
Arm/Group | Emapalumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Duration of Response
Description: as for outcome 2
Time Frame: Up to 1 year after last emapalumab administration
Population: Since the study was prematurely terminated, no data was collected for the secondary efficacy endpoints.
Arm/Group | Emapalumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Hemophagocytic Lymphohistiocytosis Relapse
Description: as for outcome 2
Time Frame: Up to 1 year after last emapalumab administration
Population: Since the study was prematurely terminated, no data was collected for the secondary efficacy endpoints.
Arm/Group | Emapalumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Incidence, Severity, Causality and Outcomes of Serious Adverse Events and Non-serious Adverse Events
Description: as for outcome 2
Time Frame: Up to 1 year after last emapalumab administration
Population: Since the study was prematurely terminated, no data was collected for the secondary safety endpoints.
Arm/Group | Emapalumab
Number analyzed (Participants) | 0

9. Secondary Outcome: Serum Concentrations of Emapalumab
Description: as for outcome 2
Time Frame: Up to 1 year after last emapalumab administration
Population: Since the study was prematurely terminated, no data was collected for the secondary Pharmacokinetic endpoints.
Arm/Group | Emapalumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Serum Biomarker Levels
Description: Levels of interferon-gamma, C-X-C chemokine ligand 9, soluble CD25, interleukin-6.
Time Frame: Up to 1 year after last emapalumab administration
Population: Since the study was prematurely terminated, no data was collected for the secondary Pharmacodynamic endpoints.
Arm/Group | Emapalumab
Number analyzed (Participants) | 0

11. Secondary Outcome: Incidence of Anti-Drug Antibodies Against Emapalumab
Description: as for outcome 2
Time Frame: Up to 1 year after last emapalumab administration
Population: Since the study was prematurely terminated, no data was collected for the secondary Pharmacodynamic endpoints.
Arm/Group | Emapalumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) reported from the first emapalumab administration up to and including Day+60 study visit were recorded, approximately 13 months.
Description: The All Treated analysis set included all patients who received at least 1 dose or 1 incomplete dose of emapalumab. Only TEAEs are reported.
Arm/Group | Emapalumab
All-Cause Mortality (participants affected / at risk) | 4/7
Serious Adverse Events (participants affected / at risk) | 5/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emapalumab (N=7)
Acute myeloid leukaemia (Blood and lymphatic system disorders) | 1 (1) — Progression of pre-existing condition
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Lymphoma (Blood and lymphatic system disorders) | 1 (1) — Progression of pre-existing condition
Bacteramia (Infections and infestations) | 1 (1)
Cytomegalovirus hepatitis (Infections and infestations) | 1 (1)
Fungaemia (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Human herpesvirus 6 encephalitis (Infections and infestations) | 1 (1)
Perineal abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emapalumab (N=7)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Lip disorder (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Escherichia bacteramia (Infections and infestations) | 1 (1)
Fungaemia (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Blood osmolarity increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Troponin T increased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Confusional state (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 2 (2)
Ajustment disorder with depressed mood (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin laceration (Skin and subcutaneous tissue disorders) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Dental disorder prophylaxis (Surgical and medical procedures) | 1 (1)
Penile haemorrhage (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Since the study was prematurely terminated, and considering the low number of patients enrolled, no analysis related to primary and secondary efficacy endpoints and no Pharmacokinetic and Pharmacodynamic summary statistics were performed. Accordingly, no conclusion on the efficacy of emapalumab on this patient population could be withdrawn from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT03985423/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT03985423/SAP_001.pdf